CLINICAL TRIAL: NCT03973567
Title: Magnetic Resonance Imaging Study of Antidepressants in the Treatment of Refractory Functional Dyspepsia
Brief Title: MRI Study of Antidepressants in the Treatment of Refractory Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-042
Record Dates: First submitted 2019-05-28; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Therapeutic Mechanism of Antidepressants for Refractory FD
Keywords: antidepressants; refractory functional dyspepsia; resting fMRI
MeSH Terms: interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Antidepressive Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- refractory FD patients using antidepressants (Experimental): Sixty FD patients who met the criteria were selected as the experimental group after more than two kinds of treatment, including acid-making, proton pump inhibitors (PPI), motivation and anti-Helicobacter pylori（HP） treatment, including 30 in the conventional treatment group and 30 in the combined antidepressant treatment group.
  Interventions: Drug: selective serotonin reuptake inhibitor (SSRI) or serotonin noradrenaline reuptake inhibitor (SNRI) antidepressants
- refractory FD patienTS using conventional treatment (Placebo Comparator): Sixty FD patients who met the criteria were selected as the experimental group after more than two kinds of treatment, including acid-making, PPI, motivation and anti-HP treatment, including 30 in the conventional treatment group and 30 in the combined antidepressant treatment group.
  Interventions: Other: conventional therapy
- normal control (No Intervention): Age, sex and education matched, right-handed 30 normal people.

INTERVENTIONS:
Drug: selective serotonin reuptake inhibitor (SSRI) or serotonin noradrenaline reuptake inhibitor (SNRI) antidepressants — On the basis of routine treatment for 8-12 weeks, according to the characteristics of symptoms, a combination of SSRI or SNRI antidepressant drugs was given for 12 weeks.
  Arms: refractory FD patients using antidepressants
Other: conventional therapy — Anti-HP, acid suppression, gastrointestinal motility regulation, etc.
  Arms: refractory FD patienTS using conventional treatment

SUMMARY:
In this study, diffusion tensor imaging（DTI）technique was used to evaluate the brain microstructures and connective white matter microstructures in patients with refractory FD, resting fMRI was used to evaluate the functional connectivity between hemispheres, and neuroimaging changes after antidepressant intervention were observed to explore the activation patterns of resting brain homeostasis-receptive network areas in patients with refractory FD. We aimed to explore microstructure of white matter and gray matter and functional connectivity between hemispheres to explain the therapeutic mechanism of antidepressants.

DETAILED DESCRIPTION:
In this study, functional magnetic resonance imaging (fMRI) was used to investigate the abnormal activation patterns of brain regions in patients with refractory FD in resting state, and to observe the changes of brain functions after antidepressant treatment, in order to find scientific evidence for exploring the etiology, neuropathological mechanism and the mechanism of antidepressant treatment of refractory FD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old, meeting the criteria for inclusion of refractory FD
* HP infection negative
* Right handedness

Exclusion Criteria:

* Antidepressant drug allergists
* History of gastroduodenal surgery;
* Researchers judged suicidal ideation.
* Women in pregnancy or lactation.
* Patients with uncorrected narrow angle glaucoma.
* There was a history of epileptic seizures.
* suffering from any serious or unstable medical disease or disease.
* Addiction to illicit drugs or alcohol and unwillingness to discontinue use during the study period.
* Patients can't express their complaints correctly and can't cooperate with the researcher.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Nepean Dyspepsia Index | Change from Baseline at 12th week
  Evaluation of digestive tract symptoms

SECONDARY OUTCOMES:
Zung Self-Rating Anxiety Scale | Change from Baseline at 12th week
  It is a scale measures anxiety level of patients including 20 items, and total score ranges from 20 to 80. Higher values represent a worse outcome.
Zung Self-Rating Depression Scale | Change from Baseline at 12th week
  It is a scale measures depression level of patients including 20 items, and total score ranges from 20 to 80. Higher values represent a worse outcome.
The Pittsburgh Sleep Quality Index | Change from Baseline at 12th week
  Assessment of Sleep Status
quality of life survey questionnaire | Change from Baseline at 12th week
  Assessment of quality of life
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 3 years
  Record any adverse events during treatment
Functional magnetic resonance imaging | baseline and 12th week
  assesses brain microstructures and connective white matter microstructures, and assesses functional connectivity between hemispheres

CONTACTS AND LOCATIONS:
Overall Officials: Yiping Chen, PHD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No